CLINICAL TRIAL: NCT04215913
Title: Integrative Analysis of Pulmonary Sarcomatoid Carcinoma (PSC)
Acronym: PSC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: The Affiliated Tumor Hospital of Nantong University, Nantong, Jiangsu Province, China (Other); Anhui Medical University (Other)
Responsible Party: Principal Investigator, Da Fu, Professor, Shanghai 10th People's Hospital
Other Study IDs: 2019-FD52Rainy-PSC; FD52Rainy (Registry Identifier: PSC)
Record Dates: First submitted 2019-12-29; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Lung Cancer
Keywords: PSC; Integrative Analysis; IHC; WES; RNA sequencing
MeSH Terms: conditions — Lung Neoplasms | interventions — DNA

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal lung tissue: Normal lung tissue from PSC patients
  Interventions: Other: The investigators will extract total protein, DNA and RNA from PSC patients.
- PSC tissues: PSC tissues from PSC patients
  Interventions: Other: The investigators will extract total protein, DNA and RNA from PSC patients.
- Metastasis tissues: Metastasis tissues from PSC patients
  Interventions: Other: The investigators will extract total protein, DNA and RNA from PSC patients.

INTERVENTIONS:
Other: The investigators will extract total protein, DNA and RNA from PSC patients. — The investigators will extract total protein, DNA and RNA from PSC patients.

SUMMARY:
Integrative Analysis of pulmonary sarcomatoid carcinoma (PSC)

DETAILED DESCRIPTION:
The investigators will analyzed proteomes of paired normal lung tissues and pulmonary sarcomatoid carcinoma with or without metastasis, sequenced transcriptomes, perform whole exome sequencing, and single nucleotide polymorphism (SNP) array profiling for triplets, each comprising normal lung tissue, primary pulmonary sarcomatoid carcinoma, and its synchronous matched metastasis, as well as analyzed genomics of lung cancer characterized previously by The Cancer Genome Atlas (TCGA) to conduct integrated proteogenomic analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 70 years with histologically proven LCLC
* No severe major organ dysfunction
* World Health Organization (WHO) performance status of 0 or 1
* No prior cancer chemotherapy

Exclusion Criteria:

* Age ≥ 70
* Severe major organ dysfunction
* WHO performance status of >1
* Prior cancer chemotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary sarcomatoid carcinoma
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-12-30 (Estimated); Primary Completion 2025-12-24 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
10 years overall survival | 10 years overall survival
  10 years overall survival

SECONDARY OUTCOMES:
10 years disease-free survival | 10 years disease-free survival
  10 years disease-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Da Fu, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Result] Boland JM, Mansfield AS, Roden AC. Pulmonary sarcomatoid carcinoma-a new hope. Ann Oncol. 2017 Jul 1;28(7):1417-1418. doi: 10.1093/annonc/mdx276. No abstract available. PMID 28637281